CLINICAL TRIAL: NCT00485017
Title: A Phase II Randomized, Double-Blind, Double-Dummy, Parallel Group, Placebo Controlled Study of THR-4109 in Obese Subjects
Brief Title: Efficacy and Safety of THR-4109 in Obese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theracos (Industry)
Collaborators: TFS Trial Form Support (Industry)
Responsible Party: Dr. E. Amento, President and CEO, Theracos, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: THR-4109-C-302
Record Dates: First submitted 2007-06-08; First posted 2007-06-12 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Obesity
Keywords: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): THR-4109: 115 mg orally in am, 115 mg orally in pm for 24 weeks
  Interventions: Drug: THR-4109
- 2 (Experimental): THR-4109: 100 mg orally in am, 100 mg orally in pm for 24 weeks
  Interventions: Drug: THR-4109
- 3 (Experimental): THR-4109: 15 mg orally in am, 15 mg orally in pm for 24 weeks
  Interventions: Drug: THR-4109
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: THR-4109 — THR-4109 maximum dose in study is 115 mg via oral capsule daily in a.m. and 115 mg via oral capsule daily in p.m. for 24 weeks
  Arms: 1; 2; 3
Drug: Placebo — Oral capsules daily in a.m. and in p.m. for 24 weeks
  Arms: 4

SUMMARY:
The purpose of this study is to evaluate the safety and effect of THR-4109 on weight loss in obese subjects over a 24-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* 30 to 60 years of age
* Body mass index between 30 and 40 kg/m2
* Women of child bearing potential with a negative pregnancy test prior to entry and who agree to use an acceptable method of contraception throughout the study
* Able and willing to give written informed consent

Exclusion Criteria:

* Weight loss of more than 3 kg in the previous 3 months
* Current or previous use (within 3 months) of medications that influence weight
* Known endocrine origin for obesity, such as hypothyroidism and Cushing's syndrome
* Current or history of eating disorder such as bulimia, anorexia nervosa, binge eating or laxative abuse
* Current serious/unstable medical condition
* Current pharmacologically treated diabetes or fasting plasma glucose ≥ 126 mg/dL

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline weight | 24 weeks

SECONDARY OUTCOMES:
Proportion of subjects who achieve weight loss of at least 5% and at least 10% of baseline body weight | 24 weeks
Serum lipids, waist circumference, fasting plasma glucose and blood pressure | 24 weeks
Safety and tolerability of THR-4109 | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Natalie J Warner, MD, Study Director — Theracos, Inc.
Locations (20):
- Russia (17):
  - Investigational Site #62, Arkhangelsk
  - Investigational Site #61, Moscow
  - Investigational Site #51, Moscow
  - Investigational Site #60, Moscow
  - Investigational Site #57, Moscow
  - Investigational Site #50, Moscow
  - Investigational Site #54, Moscow
  - Investigational Site #63, Saint Petersburg
  - Investigational Site #67, Saint Petersburg
  - Investigational Site #53, Saint Petersburg
  - Investigational Site #66, Saint Petersburg
  - Investigational Site #59, Saint Petersburg
  - Investigational Site #65, Saint Petersburg
  - Investigational Site #55, Saint Petersburg
  - Investigational Site #58, Saint Petersburg
  - Investigational Site #64, Saint Petersburg
  - Investigational Site #56, Saratov
- Sweden (3):
  - Investigational Site #12, Dalby
  - Investigational Site #11, Gothenburg
  - Investigational Site #13, Malmo